CLINICAL TRIAL: NCT02421042
Title: A Pharmacokinetic and Safety Study of E7080 in Subjects With Mild (10 mg), Moderate (10 mg), and Severe Hepatic Impairment (5 mg) and Normal Hepatic Function (10 mg)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-006
Record Dates: First submitted 2014-07-22; First posted 2015-04-20 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Hepatic Impairment; Hepatic Function
Keywords: Hepatic Impairment; Hepatic Function
MeSH Terms: interventions — lenvatinib

ARMS (1):
- Lenvatinib (Experimental): Subjects determined to be eligible for the protocol will receive either a 5- or 10-mg single oral dose of lenvatinib on Day 1, depending on their hepatic status [Mild (10 mg), Moderate (10 mg), and Severe Hepatic Impairment (5 mg) and Normal Hepatic Function (10 mg)].
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — 5- or 10-mg single oral dose of E7080, depending on their hepatic status [Mild (10 mg), Moderate (10 mg), and Severe Hepatic Impairment (5 mg) and Normal Hepatic Function (10 mg)].
  Other Names: E7080

SUMMARY:
This is a multi-center, open-label, non-randomized, single-dose, sequential-cohort study in subjects with varying degrees of hepatic impairment, classified according to the Child-Pugh system, who will be matched with normal healthy subjects as controls.

DETAILED DESCRIPTION:
This is a multi-center, open-label, non-randomized, single-dose, sequential-cohort study in subjects with varying degrees of hepatic impairment, classified according to the Child-Pugh system, who will be matched with normal healthy subjects as controls. The study will be conducted in two phases: Pretreatment and Treatment. The Pretreatment Phase will have two periods: Screening and Baseline. The study will enroll a sufficient number of subjects so that at least 24 subjects complete the study. This will include six subjects with mild hepatic impairment (Group 1), six subjects with moderate hepatic impairment (Group 2), four to six subjects with severe hepatic impairment (Group 3), and eight subjects with normal hepatic function (Group 4). Potential study subjects with hepatic impairment (Groups 1, 2, and 3) and those with normal hepatic function (Group 4) will first be screened for study entry. Group 1, 2, and 3 subjects will be enrolled sequentially into the study first. The Group 4 normal healthy subjects will be enrolled following enrollment of all of the hepatic impairment subjects. Subjects determined to be eligible for the protocol will receive either a 5- or 10-mg single oral dose of lenvatinib on Day 1, depending on their hepatic status. Subjects will be discharged from the unit on Day 17 (+/- 2 days) after all study discharge procedures have been completed.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet all of the following criteria to be included in this study:

1. Male or female subjects aged 18 to 70, inclusive
2. BMI greater than or equal to 18 to lesser than or equal to 35 kg/m2, inclusive
3. Non-smokers and smokers who smoke no more than 10 cigarettes per day
4. All females must have a negative serum beta human chorionic gonadotropin (B-hCG) test result and a negative urine pregnancy test result at Screening and Baseline. Females of childbearing potential must agree to use a highly effective method of contraception (e.g., abstinence, an intrauterine device [IUD], a barrier method such as a condom plus spermicide or condom plus diaphragm with spermicide, a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. The only subjects who will be exempt from this requirement are postmenopausal females (defined as at least 12 months' consecutive amenorrhea, in the appropriate age group, without other known or suspected primary cause) or subjects who have been sterilized surgically or who are otherwise proven sterile (i.e., bilateral tubal ligation with surgery at least 1 month prior to dosing, hysterectomy, or bilateral oophorectomy with surgery at least 1 month prior to dosing). All women who are of reproductive potential and who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
5. Male subjects who are not abstinent or have not undergone a successful vasectomy, who are partners of women of childbearing potential, must use, or their partners must use, a highly effective method of contraception (e.g., condom plus spermicide, condom plus diaphragm with spermicide, IUD) starting for at least one menstrual cycle prior to starting study drug(s) and throughout the entire study period and for 30 days (longer if appropriate) after the last dose of study drug.
6. Voluntarily provide written informed consent prior to any study procedures
7. Are willing and able to comply with all aspects of the protocol for the duration of the study.

Additionally, for subjects with hepatic impairment (based on the Child-Pugh classification system), the following key inclusion criteria will apply:

1. Subjects must have a diagnosis of liver cirrhosis that has been stable, without any change in disease status, for 60 days prior to study screening, as determined by the investigator.
2. Subjects must have a platelet count greater than 30,000 cells/mm3; if platelet count is lesser than 30,000 cells/mm3, the subject may be enrolled with joint approval of the principal investigator (PI) and medical monitor based on subject history and stability.
3. Subjects must have no history of clinically relevant disease or condition (e.g., significant cardiac or renal dysfunction, diseases of the gastrointestinal tract or conditions which may impact drug absorption), as determined by the investigator.
4. Subjects must have a total score on the Child-Pugh classification system between 5 and 6 (Group 1, mild impairment), 7 to 9 (Group 2, moderate impairment), and 10 to 15 (Group 3, severe impairment).
5. Subjects with a history of Type I or Type II diabetes are permissible, providing that, in the opinion of the investigator, they have stable disease. Subjects receiving insulin therapy are permissible provided that they have been on a stable treatment for at least 2 weeks prior to study enrollment and continuing through the study.

Exclusion Criteria:

All subjects who meet any of the following criteria will be excluded from participation in the study:

1. Use of any new medication, including multi-vitamins, or an investigational drug within 14 days prior to the drug administration, or within five times the elimination half-life, whichever is longest, except combined oral contraceptives and occasional use of paracetamol or ibuprofen within 14 days and Vitamin K supplements and thiamine for hepatic impairment subjects; any local anesthetic within 3 days before study drug administration. Current over-the-counter (OTC) and prescription medication use is permitted, but must be stable and consistent for at least 14 days prior to screening and throughout the study treatment period.
2. Positive human immunodeficiency virus (HIV) screening test
3. QTc interval calculated by Fridericia's formula (QTcF) greater than 480 ms at screening or baseline
4. Presence of acute active liver disease or acute liver injury as indicated by (1) an abnormal liver function test, or (2) clinical and/or laboratory signs of acute, active hepatitis A, B, and/or C. Subjects with stable, chronic, active hepatitis B or C may be enrolled if the investigator deems them to be appropriate.

Additionally normal healthy subjects who meet any of the following criteria will be excluded from participation in the study:

1. Presence of clinically significant illness requiring treatment
2. History of gastrointestinal surgery (cholecystectomy and appendectomy are, however, permitted)
3. History of significant drug, food, or seasonal allergies
4. Weight change during the Pretreatment Phase
5. Significant findings revealed by the history, physical or clinical laboratory testing
6. Alcohol misuse
7. Caffeine intake within 72 hours of lenvatinib administration
8. Participation in another clinical trial within 4 weeks of lenvatinib administration
9. Receipt or donation of blood or blood products within 4 to 8 weeks of lenvatinib administration
10. Engagement in strenuous exercise
11. Unwillingness to abide by the study requirements, or, in the opinion of the investigator, unlikely to complete the study.

Additionally subjects with hepatic impairment who meet any of the following criteria will be excluded from participation in the study:

1. Subjects who have a history of hepatic transplant, systemic lupus erythematosus, or hepatic coma within 2 months prior to the Screening Period
2. Subjects who are receiving or have received treatment with interferon or pegylated interferon within the past 60 days
3. Subjects who have encephalopathy greater than Grade 2, sepsis, or gastrointestinal bleeding within 1 month before the Screening Period; esophageal varices greater than Grade 2, acute hepatic failure of any etiology, history of surgical portosystemic shunt, renal impairment (creatinine clearance lesser than 50 mL/min according to the Cockcroft-Gault formula), and rapidly deteriorating hepatic function indicated recently by clinical/laboratory signs of hepatic impairment within 2 months prior to the Screening Period.
4. Subjects who have significant acute, new onset illness within 2 weeks prior to study drug administration
5. In addition to the Key Exclusion Criteria above for all subjects, standard exclusion criteria for subjects with hepatic impairment in Phase 1 studies will be used. These include the presence of clinically significant illness requiring treatment where said illness is unrelated to their hepatitis, history of gastrointestinal surgery (cholecystectomy and appendectomy are, however, permitted); history of significant drug, food, or seasonal allergies; weight change during the PreTreatment Phase; significant findings revealed by the history, physical, or clinical laboratory testing where said findings are unrelated to the subject's hepatitis, alcohol misuse, or caffeine intake within 72 hours of E7080 administration; participation in another clinical trial within 4 weeks of lenvatinib administration; receipt or donation of blood or blood products within 4 to 8 weeks of lenvatinib administration; engagement in strenuous exercise; unwillingness to abide by the study requirements; or, in the opinion of the investigator, unlikely to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of lenvatinib: Cmax | 336 hours post study drug administration
  Plasma concentrations of lenvatinib (free and total) and its metabolites, M1, M2, M3, and M5, (total) and urine concentrations of lenvatinib (total) and its metabolites, M1, M2, M3, and M5, (total) will be assessed.
Pharmacokinetics of lenvatinib: AUC(0-t) | 336 hours post study drug administration
  Plasma concentrations of lenvatinib (free and total) and its metabolites, M1, M2, M3, and M5, (total) and urine concentrations of lenvatinib (total) and its metabolites, M1, M2, M3, and M5, (total) will be assessed.
Pharmacokinetics of lenvatinib: AUC(0-inf) | 336 hours post study drug administration
  Plasma concentrations of lenvatinib (free and total) and its metabolites, M1, M2, M3, and M5, (total) and urine concentrations of lenvatinib (total) and its metabolites, M1, M2, M3, and M5, (total) will be assessed.
Safety of lenvatinib as assessed by Vital Signs | Screening, Baseline and Treatment [upto Study discharge (17 days plus or minus 2 days)]

SECONDARY OUTCOMES:
Safety of lenvatinib as assessed by Adverse Events/Serious Adverse Events | Screening, Baseline and Treatment [upto Study discharge (17 days plus or minus 2 days)]
Safety of lenvatinib as assessed by Laboratory Values | Screening, Baseline and Treatment [upto Study discharge (17 days plus or minus 2 days)]
Safety of lenvatinib as assessed by ECGs | Screening, Baseline and Treatment [upto Study discharge (17 days plus or minus 2 days)]

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Miami, Florida
  - Orlando, Florida
  - Minneapolis, Minnesota
  - Knoxville, Tennessee